CLINICAL TRIAL: NCT00126737
Title: Home-Based Exercise and Weight Control Program for Pain Control in Overweight Elderly With Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: E2920-R
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Diseases; Obesity; Osteoarthritis; Pain
Keywords: Elderly; Exercise; lean body mass; muscle strength; Nutrition program; Pain control; stair climb; walking distance; weight loss
MeSH Terms: conditions — Chronic Disease; Obesity; Osteoarthritis; Pain; Motor Activity; Agnosia; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Active Comparator): Group assigned to both a Weight Control Nutritional Program and home-based exercise program (Ex+WC).
  Interventions: Other: Weight Control Nutritional Program; Other: Home-based exercise program
- Arm 2 (Active Comparator): Group assigned to a Weight Control Nutritional Program (WC).
  Interventions: Other: Weight Control Nutritional Program
- Arm 3 (Active Comparator): Group assigned to a home-based exercise program (Ex).
  Interventions: Other: Home-based exercise program
- Arm 4 (No Intervention): Usual care and non- specific health information (C).

INTERVENTIONS:
Other: Weight Control Nutritional Program — a week of food diary and information about dietary fat intake and proper proportions of vegetables.
  Other Names: pole striding walking exercise
  Arms: Arm 1; Arm 2
Other: Home-based exercise program — 24 week home-based exercise program encompassed aerobic exercises, isometric and isotonic exercises, and stretching exercises.
  Arms: Arm 1; Arm 3

SUMMARY:
The purpose of this study is to determine whether a home-based exercise and weight control program applied to elderly overweight individuals with painful osteoarthritis of the knee, would result in pain reduction.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common chronic disease in the United States (U.S.). Arthritis is a leading chronic illness among older adults in the U.S. Approximately 40% of individuals above 60 yr of age have OA of the knee. The primary objective of the proposed study is to determine whether individuals who are overweight with OA of the knee and who complete a 24-week home-based exercise program combined with a weight control intervention program will report significantly less pain (as measured by the WOMAC) than volunteers who participate in home-based exercise (Ex) only, weight control intervention (WC) only, or standard clinical care (C). The secondary objectives of the proposed research are to determine whether overweight individuals with OA of the knee who complete the Ex+WC program, when compared to subjects who are randomly assigned to a E, WC or C groups, demonstrate significant improvement in the following health risk profile variables: (a) improved physical function (measured by the Functional Performance Inventory), (b) improved capacity to perform stair climbing and descending, (c) improved strength, (d) increased lean body mass, (e) increase in physical activity at home (measured by pedometer step count). The proposed clinical trial will utilize a prospective, randomized two by two factorial design. Descriptive and ancova statistical method will be applied for data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Male & female 50 years old
* Diagnosis of osteoarthritis by American College of Rheumatology criteria
* Knee radiographs of Kellgren and Lawrence grade 2-4
* American Arthritis Association functional class 1-3
* Body mass index of 27

Exclusion Criteria:

* Knee arthritis which did not meet American College of Rheumatology (ACR) OA criteria
* Unable to engage in exercise or follow instruction
* Limited shoulder range of motion

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2002-10; Primary Completion 2008-02 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elly Budiman-Mak, MS MPH MD, Principal Investigator — Edward Hines Jr. VA Hospital
Locations (1):
- Edward Hines, Jr. VA Hospital, Hines, Illinois, United States

REFERENCES:
- [Result] Collins E, O'Connell S, Jelinek C, Miskevics S, Budiman-Mak E. Evaluation of psychometric properties of Walking Impairment Questionnaire in overweight patients with osteoarthritis of knee. J Rehabil Res Dev. 2008;45(4):559-66. doi: 10.1682/jrrd.2007.04.0053. PMID 18712641
- [Result] Wolf S, Foley S, Budiman-Mak E, Moritz T, O'Connell S, Jelinek C, Collins EG. Predictors of weight loss in overweight veterans with knee osteoarthritis who participated in a clinical trial. J Rehabil Res Dev. 2010;47(3):171-81. doi: 10.1682/jrrd.2009.08.0136. PMID 20665344
- [Result] Possley D, Budiman-Mak E, O'Connell S, Jelinek C, Collins EG. Relationship between depression and functional measures in overweight and obese persons with osteoarthritis of the knee. J Rehabil Res Dev. 2009;46(9):1091-8. doi: 10.1682/jrrd.2009.03.0024. PMID 20437315

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study sample was recruited from the general medicine and arthritis clinics of VA Hospital Hines, Illinois, and several non-VA affiliated community-based clinics.
Pre-assignment Details: 143 subjects were screened for eligibility in the study. 33 subjects were excluded; reasons for exclusion: 7 = cardiovascular (CV) , 3 = hospitalized, 1= knee surgery, 6 = no transport, 5 = impaired cognition, 4 = spouse illness, 4= moved, and 3 = disagree with assignment/not interested. 110 subjects were then randomized.
Groups:
- Weight Control Nutritional and Home-based Exercise Program: Group assigned to both a Weight Control Nutritional Program and home-based exercise program (Ex+WC).
  Weight Control Nutritional Program: a week of food diary and information about dietary fat intake and proper proportions of vegetables Home-based exercise program: 24 week home-based exercise program encompassed aerobic exercises, isometric and isotonic exercises, and stretching exercises
- Weight Control Nutritional Program: Group assigned to a Weight Control Nutritional Program (WC).
  Weight Control Nutritional Program: a week of food diary and information about dietary fat intake and proper proportions of vegetables.
- Home-based Exercise Program: Group assigned to a home-based exercise program (Ex).
  Home-based exercise program: 24 week home-based exercise program encompassed aerobic exercises, isometric and isotonic exercises, and stretching exercises.
- Usual Care: Usual care and non-specific health information (C). No intervention.
Period: Overall Study
Arm/Group | Weight Control Nutritional and Home-based Exercise Program | Weight Control Nutritional Program | Home-based Exercise Program | Usual Care
Started | 28 | 27 | 30 | 25
Completed | 22 | 24 | 24 | 18
Not Completed | 6 | 3 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Weight Control Nutritional and Home-based Exercise Pro: Group assigned to both a Weight Control Nutritional Program and home-based exercise Program (Ex+WC).
  Weight Control Nutritional Program: a week of food diary and information about dietary fat intake and proper proportions of vegetables Home-based exercise program: 24 week home-based exercise program encompassed aerobic exercises, isometric and isotonic exercises, and stretching exercises.
- Total: Total of all reporting groups
Arm/Group | Weight Control Nutritional and Home-based Exercise Pro | Weight Control Nutritional Program | Home-based Exercise Program | Usual Care | Total
Number analyzed (Participants) | 28 | 27 | 30 | 25 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (9.6) | 66.3 (7.3) | 65.8 (7.6) | 69.5 (8.5) | 67.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 3 | 1 | 11
  Male | 23 | 25 | 27 | 24 | 99
Race/Ethnicity, Customized [Number; unit: participants]
  White | 24 | 23 | 28 | 24 | 99
  Non-white | 4 | 4 | 2 | 1 | 11
BMI at Baseline [Mean (Standard Deviation); unit: kg/m^2] | 33.8 (6.4) | 36.8 (6.2) | 34.3 (5.4) | 32.8 (5.1) | 34.4 (5.9)
Duration of OA [Mean (Standard Deviation); unit: years] — Duration of Osteoarthritis (OA) of the knee
  years | 9.1 (10.4) | 9.4 (6.0) | 11.5 (13.2) | 10.0 (9.8) | 10.0 (10.1)
Walking Distance [Mean (Standard Deviation); unit: meters] — Average distance walked in six minutes.
  meters | 414.9 (92.6) | 445.1 (125.4) | 476.9 (101.4) | 435.1 (82.4) | 443.8 (102.7)
WOMAC Function [Mean (Standard Deviation); unit: Score] — Western Ontario and McMaster University Osteoarthritis Index (WOMAC) as a full scale, it consists of pain scale, function scale, and stiffness scale. It is used to measure pain, function, and stiffness in patients with Osteoarthritis (OA) of the knee.
  We used the Function Scale only for this study. The Function Scale has 17 items, the responses are in Likert scale; namely 0=No difficulty, 1=Slight, 2=Moderate, 3= Very, 4=Extremely. The total score ranges from 0 to 68, a higher score means worse functioning. A score of 68 indicates extremely difficult in functioning.
  Score | 44.0 (11.4) | 39.2 (12.0) | 40.3 (10.6) | 44.4 (14.8) | 41.9 (12.2)
36 Items Short Form Survey Instrument (SF-36v) Mental Scale [Mean (Standard Deviation); unit: score] — The Rand Short Form-36 (SF-36). It has Physical Health and Mental Health components. Mental Health component consisted of 4 scales; they are: Vitality ( 4 items), Social functioning (2 items), Role Emotional (3 items), and Mental Health (5 items). The mental health summary measures is called the Mental health component of SF36v. It was used to measure health related quality of life. The total score ranged from 0 -100, a score of 50 is the normative average for general mental health. Lower scores correspond to worse mental health status, higher scores correspond to better mental health status.
  score | 52.1 (10.6) | 51.9 (9.8) | 48.2 (11.4) | 48.3 (11.5) | 50.1 (10.8)
SF-36v Physical Scale [Mean (Standard Deviation); unit: score] — The Rand Short Form-36 (SF-36). We used Physical Health component for self reporting of general physical health.Physical Health consists of 4 scales, Physical Function (10 items), Role Physical (4 items), Bodily Pain (2 items), General Health (5 items). The Physical Health component is a summary measure of scales, and the scores ranges from 0 to 100, a score of 50 is the normative average of general physical health. Lower scores correspond to worse physical health status, higher scores correspond to better physical health status.
  score | 34.7 (7.8) | 41.1 (7.2) | 35.7 (8.2) | 36.4 (9.0) | 36.9 (8.3)
Stair Total (climb, descend) [Mean (Standard Deviation); unit: stairs] — Total amount of stairs climbed and descended for three minutes. Subjects climbed four steps up and descended four steps down.
  stairs | 167.7 (52.5) | 181.0 (53.2) | 182.9 (54.1) | 171.7 (52.8) | 176.0 (52.8)
Married [Number; unit: participants]
  Married | 13 | 18 | 20 | 16 | 67
  Not-Married | 15 | 9 | 10 | 9 | 43

OUTCOME MEASURES:

1. Primary Outcome: WOMAC Function
Description: Western Ontario and McMaster University Osteoarthritis Index (WOMAC) is used to measure pain, function, and stiffness in patients with OA of the knee. At 24 weeks post-baseline, the average change in score was measured. We used the Function Scale only for this study. The Function Scale has 17 items, the responses are in Likert scale; namely 0=No difficulty, 1=Slight, 2=Moderate, 3= Very, 4=Extremely. The total score ranges from 0 to 68, a higher score means worse functioning. A score of 68 indicates extremely difficult in functioning.
Time Frame: Between Base-line and 24 weeks
Population: There are discrepancies in the numbers of participants being analyzed due to incomplete data collection. the disprepancies are in the following groups: 2 in Weight control Nutritional and home -based Exercise program, 3 in Weight Control Nutritional Program, 1 in Home-based exercise program and 1 in Usual Care.
Measure: Mean (95% Confidence Interval); unit: Change in Score
Arm/Group | Weight Control Nutritional and Home-based Exercise Pro | Weight Control Nutritional Program | Home-based Exercise Program | Usual Care
Number analyzed (Participants) | 20 | 21 | 23 | 17
Change in Score | -10.4 [-15.4 to -5.0] | -4.8 [-8.7 to -0.9] | -4.9 [-7.8 to -2.0] | -1.6 [-9.0 to 5.8]
Statistical Analysis 1: Comparison: Weight Control Nutritional and Home-based Exercise Pro vs Usual Care; Test type: Superiority or Other; p = 0.0129, ANCOVA; Co-variates entered into the model were BMI and WOMAC function subscale; Mean Difference (Final Values) = -6.395, 95% CI 2-sided [-11.41 to -1.38]
Statistical Analysis 2: Comparison: Weight Control Nutritional Program vs Usual Care; Test type: Superiority or Other; p = 0.0535, ANCOVA; Covariates entered into the model were BMI and WOMAC function; Mean Difference (Final Values) = -5.174, 95% CI 2-sided [-10.43 to 0.079]

2. Primary Outcome: Physical Scale SF-36v
Description: The Rand Short Form-36 (SF-36) was used to measure health related quality of life (i.e. physical health). The average change in score 24 weeks post-baseline was measured. Physical Health consists of 4 scales, Physical Function (10 items), Role Physical (4 items), Bodily Pain (2 items), General Health (5 items). The Physical Health component is a summary measure of scales, and the scores ranges from 0 to 100, a score of 50 is the normative average of general health. Lower scores correspond to worse physical health, higher scores correspond to better physical health.
Time Frame: Between Base-line and 24 weeks
Population: There are discrepancies in the numbers of participants being analyzed due to incomplete data collection. the disprepancies are in the following groups: 1 in Weight control Nutritional and home -based Exercise program, 3 in Weight Control Nutritional Program, 3 in the Usual Care.
Measure: Mean (95% Confidence Interval); unit: Change in score
Arm/Group | Weight Control Nutritional and Home-based Exercise Pro | Weight Control Nutritional Program | Home-based Exercise Program | Usual Care
Number analyzed (Participants) | 21 | 21 | 24 | 15
Change in score | 5.51 [1.38 to 9.88] | 0.56 [-2.32 to 3.44] | 3.58 [-0.83 to 8.00] | 0.34 [-4.19 to 4.88]
Statistical Analysis 1: Comparison: Weight Control Nutritional and Home-based Exercise Pro vs Usual Care; Test type: Superiority or Other; p = 0.0307, ANCOVA; Mean Difference (Final Values) = 4.545, 95% CI 2-sided [0.432 to 8.659]

3. Primary Outcome: Mental Scale SF-36v
Description: The Rand Short Form-36 (SF-36) was used to measure health related quality of life (i.e. mental health). The average change in score 24 weeks post-baseline was measured. Mental Health component consisted of 4 scales; these are the scales: Vitality ( 4 items), Social functioning (2 items), Role Emotional (3 items), and Mental Health (5 items). The mental health summary measures is called the Mental health component of SF36v. It was used to measure health related quality of life (i.e. mental health). The total score ranged from 0 to 100, a score of 50 is the normative average for general mental health. Lower scores correspond to worse mental health status, higher scores correspond to better mental health status.
Time Frame: Between Base-line and 24 weeks
Population: There are discrepancies in the numbers of participants being analyzed due to incomplete data collection. the disprepancies are in the following groups: 1 in Weight control Nutritional and home -based Exercise program, 3 in Weight Control Nutritional Program and 3 in Usual Care
Measure: Mean (95% Confidence Interval); unit: Change in Score
Groups:
- Weight Control Nutritional and Home-based Exercise pr: Group assigned to both a Weight Control Nutritional Program and home-based exercise program (Ex+WC).
  Weight Control Nutritional Program: a week of food diary and information about dietary fat intake and proper proportions of vegetables Home-based exercise program: 24 week home-based exercise program encompassed aerobic exercises, isometric and isotonic exercises, and stretching exercises.
Arm/Group | Weight Control Nutritional and Home-based Exercise pr | Weight Control Nutritional Program | Home-based Exercise Program | Usual Care
Number analyzed (Participants) | 21 | 21 | 24 | 15
Change in Score | 0.28 [-3.57 to 4.12] | 2.62 [-1.11 to 6.35] | -0.23 [-3.25 to 2.80] | -2.64 [-8.16 to 2.88]

4. Secondary Outcome: Walking Distance
Description: Average distance walked in six minutes. The average change in distance walked (meters) 24 weeks post-baseline was measured.
Time Frame: Between Base-line and 24 weeks
Population: There are discrepancies in the numbers of participants being analyzed due to incomplete data collection. the disprepancies are in the following groups: 1 in Weight control Nutritional and home -based Exercise program, 2 in Weight Control Nutritional Program.
Measure: Mean (95% Confidence Interval); unit: Change in Distance (m)
Arm/Group | Weight Control Nutritional and Home-based Exercise Pro | Weight Control Nutritional Program | Home-based Exercise Program | Usual Care
Number analyzed (Participants) | 21 | 22 | 24 | 18
Change in Distance (m) | 71.64 [46.04 to 97.24] | 17.42 [-12.40 to 47.25] | 42.08 [19.84 to 64.32] | 6.55 [-29.73 to 42.82]
Statistical Analysis 1: Comparison: Weight Control Nutritional and Home-based Exercise Pro vs Weight Control Nutritional Program; Test type: Superiority or Other; p = 0.0158, ANCOVA; Total disease (co-morbidity) as covariate was entered into the model; Mean Difference (Final Values) = 39.94, 95% CI 2-sided [7.655 to 72.215]
Statistical Analysis 2: Comparison: Weight Control Nutritional and Home-based Exercise Pro vs Usual Care; Test type: Superiority or Other; p = 0.0002, ANCOVA; Total disease (co-morbidity) as covariate was entered into the model; Mean Difference (Final Values) = 62.25, 95% CI 2-sided [29.97 to 94.54]
Statistical Analysis 3: Comparison: Home-based Exercise Program vs Usual Care; Test type: Superiority or Other; p = 0.0056, ANCOVA; Total disease (co-morbidity) as covariate was entered into the model; Mean Difference (Final Values) = 43.95, 95% CI 2-sided [12.54 to 75.36]

5. Secondary Outcome: Stair Total (Climb, Descend)
Description: Total amount of stairs climbed and descended for three minutes. Subjects climbed four steps up and descended four steps down. The average change in total number of steps 24 weeks post-baseline was measured.
Time Frame: Between Base-line and 24 Weeks
Population: There are discrepancies in the numbers of participants being analyzed due to incomplete data collection. the disprepancies are in the following groups: 2 in Weight control Nutritional and home -based Exercise program, 1 in Weight Control Nutritional Program, 1 in Home-based exercise Program and 1 in Usual Care.
Measure: Mean (95% Confidence Interval); unit: Change in Steps
Arm/Group | Weight Control Nutritional and Home-based Exercise Pro | Weight Control Nutritional Program | Home-based Exercise Program | Usual Care
Number analyzed (Participants) | 20 | 23 | 23 | 17
Change in Steps | 39.75 [28.78 to 50.72] | 23.61 [8.51 to 38.71] | 40.48 [25.82 to 55.14] | 9.06 [-10.24 to 28.36]
Statistical Analysis 1: Comparison: Weight Control Nutritional and Home-based Exercise Pro vs Usual Care; Test type: Superiority or Other; p = 0.0018, ANCOVA; Kellgren Lawrence Scale was entered into the model; Mean Difference (Final Values) = 28.129, 95% CI 2-sided [10.767 to 45.492]
Statistical Analysis 2: Comparison: Home-based Exercise Program vs Usual Care; Test type: Superiority or Other; p = 0.0024, ANCOVA; Kellgren Lawrence scale was entered into the model; Mean Difference (Final Values) = 26.71, 95% CI 2-sided [9.675 to 43.746]
Statistical Analysis 3: Comparison: Weight Control Nutritional Program vs Usual Care; Test type: Superiority or Other; p = 0.0368, ANCOVA; Kellgren Lawrence Scale was entered into the model; Mean Difference (Final Values) = 18.747, 95% CI 2-sided [1.169 to 36.325]

ADVERSE EVENTS:
Time Frame: 24 weeks.
Arm/Group | Weight Control Nutritional and Home-based Exercise Pro | Weight Control Nutritional Program | Home-based Exercise Program | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/30 | 0/25
Other Adverse Events (participants affected / at risk) | 6/28 | 3/27 | 7/30 | 6/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Control Nutritional and Home-based Exercise Pro (N=28) | Weight Control Nutritional Program (N=27) | Home-based Exercise Program (N=30) | Usual Care (N=25)
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Two subjects experienced severe knee pain from the study and decided to terminate their participation after being reviewed by the PI.
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Some participants experienced A. Fib unrelated to the study and terminated their participation.
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Some participants experienced Chronic Obstructive Pulmonary Disease (COPD) unrelated to the study and terminated their participation.
Chest Pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) — Some participants experienced chest pain unrelated to the study and terminated their participation.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Some participants developed pneumonia unrelated to the study and terminated their participation.
CAD (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Some participants developed Coronary Artery Disease unrelated to the study and terminated their participation.
Brain Abscess (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Some participants developed a brain abscess unrelated to the study and terminated their participation.
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Some participants developed confusion unrelated to the study and terminated their participation.
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Some participants developed cholecystitis unrelated to the study and terminated their participation.
Moved (Social circumstances) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Some participants moved away from the local area and decided to terminate their participation.
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Some patients developed colon cancer unrelated to the study and decided to terminate their participation.
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Some patients developed diverticulitis unrelated to the study and decided to terminate their participation.
Allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Some participants developed an allergy unrelated to the study and decided to terminate their participation.
Not Interested (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Some participants decided they were not interested in the study anymore and terminated their participation.

LIMITATIONS AND CAVEATS:
Due to the small number of females, the results may not be generalizable to females. Limitations include requirement of having good upper body strength, shoulder range, hand eye coordination, and an investment of purchasing poles of $30 per pair.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes